CLINICAL TRIAL: NCT05314933
Title: A Single/Multiple Ascending Dose Phase 1 Study Of The Safety, Tolerability, And Pharmacokinetics Of Intranasal 2-Deoxy-D-Glucose In Normal Healthy Volunteers
Brief Title: Safety and Pharmacokinetic Study of Intranasal 2-DG in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: G.ST Antivirals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2-DG-01
Record Dates: First submitted 2022-02-03; First posted 2022-04-07 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Acute Nasopharyngitis
Keywords: Virus disease; Respiratory infection; Common cold virus; Rhinovirus
MeSH Terms: conditions — Common Cold; Virus Diseases; Respiratory Tract Infections | interventions — Deoxyglucose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study drug (Active Comparator): Each subject receives either a single dose (SAD) or a multiple dose (MAD) of a 3.5% 2-Deoxyglucose as nasal spray solution.
  The starting dose for the first cohort is 3.5 mg/day up to a maximum of 84 mg/day at cohort 6.
  Interventions: Drug: 2-Deoxyglucose
- Placebo (Placebo Comparator): Each subject receives either a single (SAD) or multiple (MAD) dose of placebo. The dose for each cohort is corresponding the amount of solution needed in the verum group.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: 2-Deoxyglucose — Intranasal administration
  Other Names: 2-DG; 2-Deoxy-D-glucose
  Arms: Study drug
Other: Placebo — Intranasal administration
  Arms: Placebo

SUMMARY:
2-DG-01 is a randomized, double-blind, placebo-controlled, single and multiple ascending dose phase 1 study assessing safety, tolerability and pharmacokinetics of 2-DG in normal healthy volunteers (NHV). The safety and pharmacokinetics of 2-DG are assessed after single or multiple intranasal administrations.

DETAILED DESCRIPTION:
2-DG-01 is a randomized, placebo-controlled, double- blind single and multiple ascending dose phase 1 study in normal healthy male and female volunteers aged 18 years or older.

The primary objective of this study is to assess the clinical safety and tolerability of intranasal 2-DG in NHVs.

The secondary objective of this study is to assess the human pharmacokinetics of 2-DG.

The study is divided in two sub-parts: Part A, a single ascending dose (SAD) study of 2-DG and Part B, a multiple ascending dose (MAD) study.

Part A consists of 3 cohorts: Cohorts 1 and 2 with a randomization ratio for 2-DG to placebo of 4:1 and Cohort 3 with a randomization ratio for 2-DG to placebo of 8:2.

Part B consists of 3 cohorts: Cohort 4 with a a randomization ratio for 2-DG to placebo of 4:1 and Cohorts 5 and 6 with a randomization ratio for 2-DG to placebo of 8:2.

Cohorts 1, 2 and 4 will also be controlled by randomized intranasal application of placebo into the opposite nostril to obtain an intra-individual estimate for local tolerability. Other cohorts will receive either 2-DG or placebo into both nostrils.

Interim safety reviews are performed by a Data Monitoring Committee.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female volunteers, age ≥ 18 years old at screening
* Females must be post-menopausal (> 1 year since last menstruation)
* Able to comprehend and to give informed consent
* Able to cooperate with the investigator, to comply with the requirements of the study, and to complete the full sequence of protocol-related procedures
* Undergone full immunisation against SARS-CoV2 or status post infection with SARS-CoV2 (both as defined by the Austrian Ministry of Health)

Exclusion Criteria:

* Frequent epistaxis (equal to or greater than 1/month)
* Hypo- or anosmia
* Symptoms of rhinitis, allergy or common cold disease at screening and at study initiation
* Medical history of diabetes mellitus of any type
* Clinically relevant abnormal findings at screening
* Preceding nasal surgery or sinus surgery
* Medical history of allergic rhinitis or chronic condition of the upper or lower respiratory tract with active symptoms within 30 days prior to screening
* SARS-CoV-2 infection positive by PCR test at screening
* Vulnerable subjects as defined by GCP
* Subjects in a dependency relationship towards the investigators, e.g. as employees
* Substance abuse, mental illness, or any reason that makes it unlikely in the judgment of the investigator for the subject to be able to comply fully with study procedures
* Use of medication (including prophylactic treatments) during 2 weeks before the start of the study, which in the judgment of the investigator may adversely affect the subject's welfare or the integrity of the study's results
* Concurrent treatment with other experimental product or participation in another clinical trial with any investigational product within 30 days or 5 elimination half-lives (whichever is longer) prior to treatment start
* Scheduled vaccination appointments during the study period

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-09-27 (Actual)

PRIMARY OUTCOMES:
Adverse drug reactions (ADRs) | until 24 hours after single drug dosing
  Number of ADRs after a single dose of 2-DG assessed by type, frequency and severity of ADRs graded as per Common Terminology Criteria for Adverse Events (CTCAE).
Adverse drug reactions (ADRs) | until 168 hours after start of multiple drug dosing
  Number of ADRs after multiple doses of 2-DG assessed by type, frequency and severity of ADRs graded as per Common Terminology Criteria for Adverse Events (CTCAE).

SECONDARY OUTCOMES:
Biodistribution of a single dose of 2-DG | baseline,0.5 hours, 2 hours, 4 hours, 6 hours after single drug dosing
  Analysis of 2-DG concentrations in plasma and nasal wash samples measured by LC-MS (µg/ml).
Biodistribution of multiple doses of 2-DG | baseline, 12 hours, 15 hours, 24 hours, 72 hours, 168 hours after start of multiple drug dosing
  Analysis of 2-DG concentrations in plasma and nasal wash samples measured by LC-MS (µg/ml).
Local tolerability of a single dose of 2-DG | baseline, 6 hours, 24 hours after single drug dosing
  Abnormal physical examination findings in the nasal cavity (type, frequency, severity of medical abnormalities, scoring of self-reported symptoms).
Local tolerability of multiple doses of 2-DG | baseline, 3 hours, 12 hours, 24 hours after start of multiple drug dosing
  Abnormal physical examination findings in the nasal cavity (type, frequency, severity of medical abnormalities, scoring of self-reported symptoms).
Olfactory function after a single dose of 2-DG | baseline, 24 hours after single drug dosing
  Change in olfactory capacity using sniffing sticks measured by Threshold-Discrimination-Identification score (TDI score). Minimum value = 0 , maximum value= 48. A higher score means a better outcome.
Olfactory function after multiple doses of 2-DG | baseline, 24 hours, 72 hours, 168 hours after start of multiple drug dosing
  Change in olfactory capacity using sniffing sticks measured by Threshold-Discrimination-Identification score (TDI score). Minimum value = 0 , maximum value= 48. A higher score means a better outcome.
Premature terminations due to ADRs after a single dose of 2-DG | until 24 hours after single drug dosing
  Number of premature terminations due to ADRs that are assessed by type, frequency and severity graded as per Common Terminology Criteria for Adverse Events (CTCAE).
Premature terminations due to ADRs after multiple doses of 2-DG | until 168 hours after start of multiple drug dosing
  Number of premature terminations due to ADRs that are assessed by type, frequency and severity graded as per Common Terminology Criteria for Adverse Events (CTCAE).
Adverse events after single dose 2-DG | until 24 hours after single drug dosing
  Number of AEs assessed by type, frequency and severity graded as per Common Terminology Criteria for Adverse Events (CTCAE).
Adverse events after multiple doses 2-DG | until 168 hours after start of multiple drug dosing
  Number of AEs assessed by type, frequency and severity graded as per Common Terminology Criteria for Adverse Events (CTCAE).

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bischof T, Gsoellpointner M, Miljevic KDK, Moser MM, Dizdarevic AM, Gualdoni GA, Gorki AD, Nicolodi C, Chou S, Radivojev S, Haiden N, Mueller CA, Firbas C, Jilma B, Schoergenhofer C. Safety, tolerability, and pharmacokinetics of intranasal 2-deoxy-D-glucose in normal healthy volunteers: A randomized, double-blind, placebo-controlled, single and multiple ascending dose phase 1 study. Eur J Pharm Sci. 2025 Jun 1;209:107069. doi: 10.1016/j.ejps.2025.107069. Epub 2025 Mar 16. PMID 40101848